CLINICAL TRIAL: NCT01433770
Title: Effects of Alefacept on Donor-Specific Memory in Kidney Transplant Recipients
Brief Title: Alefacept in Kidney Transplant Recipients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The drug will no longer be available in the United States.
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Principal Investigator, Donald Hricik, Professor of Medicine, Chief Division of Nephrology and Hypertension, Medical Director Transplantation Services, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 02-11-06
Record Dates: First submitted 2011-09-08; First posted 2011-09-14 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alefacept action on memory T cells (Experimental)
  Interventions: Drug: Amevive

INTERVENTIONS:
Drug: Amevive — Alefacept 15mg subcutaneous; once a week for 12 weeks
  Other Names: Alefacept

SUMMARY:
Alefacept, also known as Amevive®, is a medication approved by the Food and Drug Administration (FDA) in the United States and other countries for the treatment of psoriasis, which is a chronic inflammatory immunological skin condition that can result in chronic dry, red patches that are covered in scales. Alefacept is approved by the FDA for the treatment of psoriasis but not as an anti-rejection medication in transplant patients. It is now being tested in new kidney transplant patients as a supplement to other approved anti-rejection drugs. Alefacept will be used as an investigational drug in this study.

The reason for this study is to test whether using Alefacept will inhibit T cells, known as memory cells, using a test named ELISPOT-IFN. In patients with psoriasis, Alefacept inhibits these memory cells. If memory cells specific to your donor can be inhibited by this drug, it might prevent rejection and promote acceptance of the transplanted kidney in a unique manner.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign informed consent
* Adult (>18years) kidney-alone transplant recipient
* 6 months post-transplant
* Persistently positive donor-stimulated ELISPOT-IFN (≥30 spots/300K cells)-2 positive assays separated by at least one week
* Female subjects of child bearing potential must have a negative urine or serum pregnancy test within 7 days prior to enrollment and must agree to maintain effective birth control during the study

Exclusion Criteria:

* Baseline CD4 count <250 cells/uL
* Acute rejection episode within the 3 months prior to enrollment
* Clinically overt infection within the 3 months prior to enrollment
* History of BK polyoma viremia
* Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV)
* Subject has a current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully
* Any major illnesses/condition that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and completion of the study, or could preclude the evaluation of the subject's response

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Absolute changes in ELISPOTS, PRT (Panel Reactive T Cells), and lymphocyte subsets will be analyzed using paired t-tests to compare baseline vs 4, 8, 12, 16, and 24 weeks of follow-up | 12, 24, and 36 months

SECONDARY OUTCOMES:
The incidence of clinically overt infections will be descriptive or calculated as a simple percentage. | 12, 24, and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald E Hricik, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States